NCT : 1690/KEPK/XII/2019

: The Effect of Combination Therapy Using Li-ESWT and PDE-5 Inhibitor Compared to PDE-5 Inhibitor Alone in Patients With Erectile Dysfunction Title

Date : November 11, 2019

## **Informed Consent**

| I, the undersigned, : | |
|---|---|
| Name | i |
| Age | · |
| Address | |
| Telp. / Email | i |
| After being explained, and gi hereby, declare that : | iven the chance to question the part which I have not understand, I AGREE |
| | 1 AGREE |
| to enroll as a subject of the tr | ial entitled: |
| | herapy Using Li-ESWT and PDE-5 Inhibitor Compared to PDE-5 Alone in Patients With Erectile Dysfunction" |
| And, at any time I can withdraw | w myself from the enrollment. |
| | Surabaya, |
| | () |
| Witness 1, | Witness 2, |